CLINICAL TRIAL: NCT06266156
Title: Evaluation of The Effect of Consecutive Dental Visits on Dental Anxiety of Paediatric Patients
Status: Completed | Type: Observational
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hamit Tunc, Asst. Prof. Dr., Burdur Mehmet Akif Ersoy University
Other Study IDs: BMU-HTUNC-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Heart Rate; Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Firts Dental Visit: Dental anxiety level, heart rate and oxygen saturation of participants in first dental visit.
  Interventions: Behavioral: Score of anxiety questionnaire; Diagnostic Test: Heart rate; Diagnostic Test: Oxygen saturation
- Second dental visit: Dental anxiety level, heart rate and oxygen saturation of participants in second dental visit.
  Interventions: Behavioral: Score of anxiety questionnaire; Diagnostic Test: Heart rate; Diagnostic Test: Oxygen saturation

INTERVENTIONS:
Behavioral: Score of anxiety questionnaire — All participants were answered the dental anxiety questionnaire.
Diagnostic Test: Heart rate — All participants heart rate were measured with finger type pulse oxymeter.
Diagnostic Test: Oxygen saturation — All participants oxygen saturation were measured with finger type pulse oxymeter.

SUMMARY:
The goal of this observational study is to learn about in effect of consecutive dental visits on dental anxiety of paediatric patients.

The main question[s]it aims to answer are:

* Did the anxiety level of pediatric patients decrease in consecutive treatment sessions?
* Were there changes in the physiological parameters related to stress level of pediatric patients in consecutive treatment sessions?

Participants will fill out the questionnaire about dental anxiety in each dental treatment sessions before and after dental treatment.

Researchers will compare paeditric patients have two caries on mandibular molars to see if changes dental anxiety levels and physiological parameters such as heart rates and oxygen saturations during dental treatments in consecutive dental treatment sessions.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of consecutive dental visits on paediatric patients' dental anxiety level in 6-9 years old Turkish children with using of Abeer Children Dental Anxiety scale and physiological parameters.

Determination of Sample Size and Study Design The significance level for the sample size in the study was regulated to show an effect size of 0.83 with a power of 0.05 and 95%. The number of samples (n) was calculated as 200. However, it was decided that the total number of samples (n) would be 260 with data loss foreseen.

According to American Society of Anaesthesiologists (ASA), ASA1 and ASA2 healthy children who 6-9 years old without any learning and physical disabilities, children who don't need to emergency dental applications, children who can speak and understand Turkish, children who have dental caries that involved only dentine and enamel and were included to this study. Children with any disabilities that physical and mental or without parental consent were excluded from this study. In addition to this, children who has a systemic disease with changing the blood pressure, oxygen saturation and heart rate were excluded from this study. 260 children who met the inclusion criteria invited to the study.

Collection of Data and Study Procedure The ACDAS that including three parts as evaluation of child, dental, cognitive and 19 questions was used as a cognitive scale for this study. In the dental part of ACDAS including 13 questions, the children answered these questions using with three types of facial expressions for to show how they felt. All the answers were scored with scale of 1-3. According to the ACDAS children who have score of 26 and above were classified as anxious. The child evaluation and cognitive parts of ACDAS were answered by the paediatric dentist and child's legal guardians. The scores of ACDAS were accepted for master scores. Children were examined by the paediatric dentist as only clinical and radiographical without any dental treatment on first visit.

All participants were recorded, and their appointments were made by the dental assistant. Children were treated with topical anaesthesia (cotton with lidocaine %10 spray) followed by buccal infiltration local anaesthesia (articaine hydrochloride %4) for caries removing of one of the primary molars. The two mandibular primary molars of children were restored with compomer resin with using the rubber dam in first and second visits. All children were directed by same paediatric dentist (HT) with non-pharmacological behaviour management techniques during the dental treatments such as tell-show-do.The treatment duration was approximately 15 minutes. All participants completed to ACDAS for the two times as pre and post operative in both visits.

The objective symptoms of evaluation of dental anxiety such as oxygen saturation and heart rate were included in this study. Heart rate and oxygen saturations of each patient were measured with pulse oximeter (PC-60FL Finger Type Pulse Oxymeter, Galena, TURKEY). The heart rate and oxygen saturation were measured in 5th, 10 th and 15th minutes in first and second visits during dental procedures.

Statistical Analysis All data were analysed with SPSS 22.0 (SPSS for Windows, SPSS Inc, Chicago, IL) and GraphPad Prism software 7.0 for Windows (GraphPad Software, San Diego, California, USA). The sample size of the study was calculated with G-Power (version 3.1.9.7, Heinrich-Heine-Universität Düsseldorf, Germany). Calculation of the normality of the data was using with Kolmorognov-Simirnov test and followed by parametric tests. All data showed normal distribution. Standard deviation (SD) and mean values were shown with numerical variables. Categorical variables were shown with percentages. Two sample t-test were performed for comparing the differences between mean ACDAS score and physiological parameters of first and second visits.

ELIGIBILITY:
Inclusion Criteria:

* According to American Society of Anaesthesiologists (ASA), ASA1 and ASA2 healthy children who 6-9 years old without any learning and physical disabilities, children who don't need to emergency dental applications, children who can speak and understand Turkish, children who have dental caries that involved only dentine and enamel and were included to this study.

Exclusion Criteria:

* Children with any disabilities that physical and mental or without parental consent were excluded from this study. In addition to this, children who has a systemic disease with changing the blood pressure, oxygen saturation and heart rate were excluded from this study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-9 years who meet the inclusion criteria and needed at least two restorative dental treatments of the mandibular first primary molar were included in the study.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Determination of sample size. | Before the starting to study
  The significance level for the sample size in the study was regulated to show an effect size of 0.83 with a power of 0.05 and 95%. The number of samples (n) was calculated as 200. However, it was decided that the total number of samples (n) would be 260 with data loss foreseen.
Inviting participants to the study. | Before the starting to study
  ASA1 and ASA2 healthy children who 6-9 years old without any learning and physical disabilities, children who don't need to emergency dental applications, children who can speak and understand Turkish, children who have dental caries that involved only dentine and enamel and were included to this study. The Abeer Children Dental Anxiety Scale that including three parts as evaluation of child, dental, cognitive and 19 questions was used as a cognitive scale for this study. All the answers were scored with scale of 1-3. Children who have score of 26 and above were classified as anxious. Heart rate and oxygen saturations of each patient were measured with pulse oximeter.
Determination of dental anxiety score of participants before dental treatment in first dental session | Before the starting to dental treatment in first session.
  All participants completed The Abeer Children Dental Anxiety Scale (ACDAS) before starting treatment.The ACDAS that including three parts as evaluation of child, dental, cognitive and 19 questions was used as a cognitive scale for this study. In the dental part of ACDAS including 13 questions, the children answered these questions using with three types of facial expressions for to show how they felt. All the answers were scored with scale of 1-3. The total scores were ranging between 13 and 39. Children who have score of 26 and above were classified as anxious.
Heart rate measuring in first dental session. | Measured at the 5th, 10th and 15th minutes of dental treatment.
  The heart rate were measured in every 5 minutes during dental procedures. Total dental treatment time 15 minutes.
Oxygen saturation measuring in first dental session. | Measured at the 5th, 10th and 15th minutes of dental treatment.
  The oxygen saturation were measured in every 5 minutes during dental procedures. Total dental treatment time 15 minutes.
Determination of dental anxiety score of participants after dental treatment in first dental session | After the dental treatment in first session.
  All participants completed the dental anxiety questionnaire after treatment process.
Determination of dental anxiety score of participants before dental treatment in second dental session | Before the starting to dental treatment in second session.
  All participants completed the dental anxiety questionnaire before starting treatment.
Heart rate measuring in second dental session. | Measured at the 5th, 10th and 15th minutes of dental treatment.
  The heart rate were measured in every 5 minutes during dental procedures. Total dental treatment time 15 minutes.
Oxygen saturation measuring in second dental session. | Measured at the 5th, 10th and 15th minutes of dental treatment.
  The oxygen saturation were measured in every 5 minutes during dental procedures. Total dental treatment time 15 minutes.
Determination of dental anxiety score of participants after dental treatment in second dental session | After the dental treatment in second session.
  All participants completed the dental anxiety questionnaire after treatment process.

CONTACTS AND LOCATIONS:
Overall Officials: Hamit Tunç, Ph.D, Principal Investigator — Burdur Mehmet Akif Ersoy University Faculty of Dentistry Deparment of Paediatric Dentistry
Locations (1):
- Burdur Mehmet Akif Ersoy University Faculty of Dentistry, Burdur, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No